CLINICAL TRIAL: NCT02587871
Title: HLA-Mismatched Allogeneic Cellular Therapy (Microtransplantation) After Chemotherapy in Patients With Intermediate-Risk Acute Myeloid Leukemia < 60 Years
Brief Title: Donor Cellular Therapy After Cytarabine in Treating Patients With Intermediate-Risk Acute Myeloid Leukemia in Remission
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: PI decided not to pursue study
Sponsor: University of Southern California (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 9L-15-2; NCI-2015-01671 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 9L-15-2 (Other: USC / Norris Comprehensive Cancer Center); P30CA014089 (NIH)
Record Dates: First submitted 2015-10-23; First posted 2015-10-27 (Estimated); Last update posted 2018-11-09 (Actual); Status verified 2018-11

CONDITIONS: Adult Acute Myeloid Leukemia in Remission; Childhood Acute Myeloid Leukemia in Remission
MeSH Terms: interventions — Cytarabine; Peripheral Blood Stem Cell Transplantation; Filgrastim

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (cytarabine, G-CSF mobilized peripheral blood cells) (Experimental): Approximately 4-6 weeks after completion of induction chemotherapy, patients receive cytarabine IV over 1-3 hours BID on days -7 to -2 and G-CSF mobilized peripheral blood cells (microtransplant) IV over 15-20 minutes on day 0. Treatment repeats every 8-10 weeks for 3 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Cytarabine; Other: Laboratory Biomarker Analysis; Procedure: Peripheral Blood Stem Cell Transplantation; Biological: Therapeutic Allogeneic Lymphocytes; Biological: G-CSF mobilized peripheral blood cells

INTERVENTIONS:
Drug: Cytarabine — Given IV
  Other Names: .beta.-Cytosine arabinoside; 1-.beta.-D-Arabinofuranosyl-4-amino-2(1H)pyrimidinone; 1-.beta.-D-Arabinofuranosylcytosine; 1-Beta-D-arabinofuranosyl-4-amino-2(1H)pyrimidinone; 1-Beta-D-arabinofuranosylcytosine; 1.beta.-D-Arabinofuranosylcytosine; 2(1H)-Pyrimidinone, 4-Amino-1-beta-D-arabinofuranosyl-; 2(1H)-Pyrimidinone, 4-amino-1.beta.-D-arabinofuranosyl-; Alexan; Ara-C; ARA-cell; Arabine; Arabinofuranosylcytosine; Arabinosylcytosine; Aracytidine; Aracytin; Aracytine; Beta-Cytosine Arabinoside; CHX-3311; Cytarabinum; Cytarbel; Cytosar; Cytosar-U; Cytosine Arabinoside; Cytosine-.beta.-arabinoside; Cytosine-beta-arabinoside; Erpalfa; Starasid; Tarabine PFS; U 19920; U-19920; Udicil; WR-28453
Other: Laboratory Biomarker Analysis — Correlative studies
Procedure: Peripheral Blood Stem Cell Transplantation — Undergo microtransplant
  Other Names: PBPC transplantation; Peripheral Blood Progenitor Cell Transplantation; Peripheral Stem Cell Support; Peripheral Stem Cell Transplantation
Biological: Therapeutic Allogeneic Lymphocytes — Undergo microtransplant
  Other Names: Allogeneic Lymphocytes; Tumor-Derived Lymphocyte
Biological: G-CSF mobilized peripheral blood cells — microtransplantation
  Other Names: Filgrastim

SUMMARY:
This phase II trial studies how well donor cellular therapy after cytarabine works in treating patients with intermediate-risk acute myeloid leukemia with a decrease in or disappearance of signs and symptoms of cancer. Donor cellular therapy is a short-term transfusion of cells from a family member who is incompletely matched. The use of these partially matched white blood cells may help improve response to standard chemotherapy (cytarabine) and reduce some of the risks of infection, without a permanent transplant. Drugs used in chemotherapy, such as cytarabine, work in different ways to stop the growth of cancer cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Giving donor cellular therapy after cytarabine may kill more cancer cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To assess 2-year disease-free survival (as defined by time to death from any cause or disease relapse, whichever is earlier) for patients < 60 years of age with intermediate-risk acute myeloid leukemia (AML), in complete remission (CR) after induction chemotherapy, who receive microtransplantation, compared to patients who received consolidation chemotherapy only in a historical published comparable cohort of patients.

SECONDARY OBJECTIVES:

I. To obtain estimates of rate of relapse, treatment related mortality (TRM), all cause mortality, in the microtransplantation (MST) group and compare it with allogeneic stem cell group (historical cohort).

II. To obtain estimates of rate acute graft-versus-host disease (GVHD), chronic GVHD, time to recovery of absolute neutrophil counts and platelets in patients with intermediate risk AML receiving of chemotherapy in combination with microtransplantation.

TERTIARY OBJECTIVES:

I. Presence or absence of detectable donor chimerism post-microtransplantation until 6 months after the last infusion.

II. Characteristics of the infused cells and composition of the graft. III. Dynamics of T-cell clonality. IV. Immune cell subset analysis.

OUTLINE:

Approximately 4-6 weeks after completion of induction chemotherapy, patients receive cytarabine intravenously (IV) over 1-3 hours twice daily (BID) on days -7 to -2 and granulocyte colony stimulating factor (G-CSF) mobilized peripheral blood cells (microtransplant) IV over 15-20 minutes on day 0. Treatment repeats every 8-10 weeks for 3 courses in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at least every 3 months for 2 years.

ELIGIBILITY:
Inclusion Criteria:

* PATIENT INCLUSION CRITERIA:
* Acute myeloid leukemia-intermediate risk as defined by standard World Health Organization (WHO) criteria for AML (at least 20% blasts in the peripheral blood or bone marrow) at the time of initial diagnosis

  * Diagnosis of AML according to WHO diagnostic criteria (at least 20% blasts in the peripheral blood or bone marrow), with French-American-British (FAB) classification other than M3 (acute promyelocytic leukemia), documented by bone marrow aspiration and biopsy performed within 14 days prior to administration of 1st dose of remission induction chemotherapy
* Intermediate risk based on National Comprehensive Cancer Network (NCCN)
* In CR or complete remission with incomplete blood count recovery (CRi) after 1-2 induction chemotherapy documented by a bone marrow examination done within 2 weeks of starting cytarabine in this protocol
* Must have achieved CR/CRi with less than 2 induction regimens that contain cytarabine and anthracycline
* No 10/10 matched sibling donor available or not financially eligible for allogeneic stem cell transplantation
* Must be within 3 months from the last induction regimen at the time of starting cytarabine chemotherapy in this protocol
* Patient has at least one medically fit first- or second-degree family member expected to be human leukocyte antigen (HLA) mismatched at 2-9/10 loci; in addition, the prospective donor is willing to voluntarily donate hematopoietic stem cells and sign consent forms
* Absolute neutrophil count (ANC) > 1500, unless due to direct bone marrow involvement of disease
* Platelets > 75,000, unless due to direct bone marrow involvement of disease
* Hemoglobin > 8.0 gm/dL, transfusion allowed
* Serum creatinine < 2.0 x the upper limits of institutional normal (ULN)
* Total bilirubin < 1.5 x the upper limits of institutional normal
* Aspartate aminotransferase (AST)/alanine aminotransferase (ALT) < 2.5 x the upper limits of institutional normal (=< 5 x ULN for patients with suspected liver involvement of leukemia)
* Cardiac left ventricular ejection fraction (LVEF) > 45%
* Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1, or 2, and estimated survival of at least 3 months
* Patients must be able to understand and agree to sign an Institutional Review Board (IRB)-approved informed consent form
* Women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control) prior to study entry, for the duration of study, and for two months after study participation; should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately
* DONOR INCLUSION CRITERIA:
* Donor screening; all donors will meet the standard blood donor criteria established by the participating local blood center, American Association of Blood Banks (AABB)
* Donors will be selected from among the subject's relatives, adult children preferred
* Infectious disease testing will be done per Hemacare policy and AAAB guidelines
* Donor and intended recipient red cell type and compatibility will be determined
* Donors will be pre-selected on the basis of HLA haploidentity
* If patient is cytomegalovirus (CMV)-negative, donors who are CMV-negative will be preferred; CMV serology of the donor will be tested prior to the allogeneic cell donation; donations from CMV-positive donors to CMV-negative recipients will be given if no CMV negative donor is available, and CMV surveillance and pre-emptive treatment given as per guidelines below

Exclusion Criteria:

* PATIENT EXCLUSION CRITERIA:
* Acute promyelocytic leukemia
* High risk AML (see NCCN risk criteria)
* Low risk AML (see NCCN risk criteria)
* Fludarabine based therapy within 6 months of enrollment
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Who are pregnant and/or lactating
* Who have had non-biopsy surgery in the last 10 days
* Who have active central nervous system (CNS) disease; patients with previously treated leptomeningeal disease without evidence of remaining leukemia cells by spinal fluid will be eligible
* Patients with known active autoimmune disorder
* Patients known to be have active hepatitis B or C; (hepatitis B positive patients are allowed if they are on appropriate antiviral agents such as lamivudine)
* Patients concurrently taking the following drugs are excluded: mycophenolate, cyclosporine, prednisone > 20 mg/day, or immunosuppressive agents
* Researchers think that any life-threatening illness, condition or organ system dysfunction can damage the safety of subjects
* Failure to demonstrate adequate compliance with medical therapy and follow-up
* DONOR EXCLUSION CRITERIA:
* Personal or family history of severe sickle cell disease or variant (unless donor has tested negative); testing for the presence of hemoglobin S is not required
* Positive infectious disease test as dictated by blood collection center's standard operating procedure (SOP)
* Current uncontrolled hypertension
* Pregnant or breast-feeding
* Currently taking lithium therapy
* History of autoimmune disease

Max Age: 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2018-12-12 (Estimated); Primary Completion 2020-11-12 (Estimated); Study Completion 2022-11-12 (Estimated)

PRIMARY OUTCOMES:
Disease free survival (DFS) | Beginning of therapy to the date of death or the date of last follow-upexamination, assessed at 2 years
  The 2-year DFS will be estimated, and the corresponding 90% confidence intervals will be constructed. The data will be displayed using a Kaplan-Meir curve to plot the DFS over time. Calculate bilateral 95% confidential interval of mean difference of disease-free survival rate, and compare the lower limit of the bilateral 95% confidential interval and 15% superiority boundary value.

SECONDARY OUTCOMES:
Cumulative incidence acute GVHD, classified as clinically significant (grades 2 to 4) or severe (grades 3 to 4) | 6 months after microtransplant
  At single time point, if univariate quantitative data of the meets the normal distribution and homogeneity of variance, perform test of univariate quantitative data, otherwise, adopt the rank-sum test of corresponding design; for univariate quantitative data under multiple time points, use mixed effects model to design variance analysis with repeated measure factors.

CONTACTS AND LOCATIONS:
Overall Officials: Giridharan Ramsingh, Principal Investigator — University of Southern California
Locations (1):
- USC / Norris Comprehensive Cancer Center, Los Angeles, California, United States